CLINICAL TRIAL: NCT03170570
Title: A Prospective Study on the Efficacy and Safety of the Re-irradiation of Recurrent Cervical Cancer Within the Irradiated Field by Intensity Modulated Radiotherapy
Brief Title: the Re-irradiation of Recurrent Cervical Cancer by IMRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xin-ping Cao, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRTCC2017
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Cervical Cancer; Radiation Toxicity; Recurrent Cervical Carcinoma
Keywords: recurrent cervical cancer; re-irradiation; intensity-modulated radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Radiation Injuries | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): retreatment using intensity-modulated radiotherapy for cervical cancer patients with in-field recurrence
  Interventions: Device: intensity-modulated radiotherapy

INTERVENTIONS:
Device: intensity-modulated radiotherapy — IMRT: intensity modulated radiotherapy, Treatment schedule: 4-7 weeks, 20-35 fractions, unless the stop indications were met, treatment will continue.

SUMMARY:
this is a prospective clinical trial using intensity modulated radiotherapy（IMRT）for the treatment of cervical cancer patients with recurrent disease within the previously irradiated field. Sixty patients will be enrolled after careful selection to meet the including criteria and excluding criteria. A primary course of 36Gy will be prescribed to the recurrent site and a further 9-24Gy of dose escalation will be prescribed to the gross tumor volume in the second course according to the toxicities and the shrinkage of tumor. Weekly concurrent cisplatin of 30mg/m2 by five weeks will be administrated intravenously to the selected patients. Acute and late toxicities will be monitored and survival endpoints will be tracked with our follow-up protocol to evaluate the safety and efficacy of this approach.

DETAILED DESCRIPTION:
Introduction: Cervical cancer is the seventh most common and the eighth deadliest cancer in Chinese women. In spite of the advances in multimodality treatment regimens, there were 15-40% patients suffering from recurrence within initial irradiated field[1, 2], of which 95% recurrence occurred within 2 years and only 20% of them could be treated by salvage treatment[3-6]. there were controversies on how recurrent cervical cancer within the irradiated field should be dealt with. Surgery such as pelvic extenteration had to remove involved organs including intestine, rectum or bladder and sometimes led to severe complications and a poor quality of life. After the initial 45-50Gy irradiated to the whole pelvis, it seemed to have minimal space of further re-irradiation for recurrent disease as conventional radiotherapy was applied when considering late toxicities of organs at risk. The radiation dose for pelvic structures received will reach 45-50 Gy, almost reached the upper limits of normal tissues. For recurrent cervical cancer patients receiving retreatment by radiotherapy, the toxicity increased by 30%-56%[2] when conventional technique was applied, toxicities restricted sufficient treatments to the recurrence disease leading to a poor prognosis, which was usually less than a year [8]. IMRT has an advantage over conventional techniques because of delivering a high dose to target volume while sparing organs at risk which were previously irradiated in the primary radiotherapy. We have a five years' experience using IMRT to treat patients with recurrent disease within the previously irradiated field and most of patients showed good response and tolerable complication. According to our retrospective research (publishing), thirty-three patients made a median survival time of 14.06 months, one year overall survival was 55% and 2 year overall survival was 22%, which were better than the results of one year survival 10-20% from previous studies [8]. For further evidence, we designed this prospective clinical trial to evaluate the efficacy and safety when using intensity modulated radiotherapy to treat patients with recurrent cervical cancer within the previously irradiated field.

Methods: Sixty patients with recurrent cervical cancer within the previously irradiated field will be prospectively enrolled in this study. Only patients meeting both the including criteria and exclusion criteria will be carefully selected considering potential severe toxicities. A primary course of 36Gy will be prescribed to the recurrent site and a further 9-24Gy of dose escalation will be prescribed to the gross tumor volume in the second course according to the toxicities and the shrinkage of tumor to the irradiation. Intensity Modulated RadioTherapy (IMRT) will be chosen for dose delivery as this technique gives sufficient dose to target volume meanwhile sparing organs at risk. Weekly cisplatin of 30mg/m2 by five weeks will be administrated intravenously to the selected patients.

Outcome measurements: Toxicities will evaluated using Common Terminology Criteria for Adverse Events version 4.0 (CTCAE 4.0). Acute toxicities will be monitored weekly until one month after the completion of radiotherapy and chemotherapy. Then late toxicities will be recorded by monthly following-up. Three year's progression free survival (3y PFS) and three year's recurrence free survival(3y RFS) are the major endpoints of this study. Every three months the patients will be evaluated with necessary modalities such as physical examination, blood test, radiography, computed tomography, magnetic resonance and/or positron emission topography until three year after the last radiotherapy/chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients have provided a signed Informed Consent Form.
* Histologically confirmed cervical cancer patients after initial radiotherapy with in-field recurrence age 18-65
* Willing to have retreatment by radiotherapy
* ECOG status 0～2，Karnofsky(KPS) score ≥80
* Normal internal organ function

Exclusion Criteria:

* Having the serious cardiovascular disease or other serious complications.
* Woman in pregnancy and breast-feeding.
* Patients who had other malignant tumors in five years .
* Patients who had epilepsy.
* Patients who had infectious diseases.
* Patients who had severe side effects from previous treatment, such as intestinal disease, radiation induced pneumonia, diabetes, renal failure and hepatic failure.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
3 year progression free survival (PFS) | evaluate the response every 3 months since the completion of treatment until the progression of disease or death of patient up to 36 months
  3 year progression free survival

SECONDARY OUTCOMES:
3 year recurrence free survival ( RFS) | evaluate the response every 3 months since the completion of treatment until the recurrence of disease or death of patient up to 36 months
  3 year recurrence free survival

OTHER OUTCOMES:
3 year overall survival ( OS) | evaluate the response every 3 months since the completion of treatment until the death of patient up to 36 months
  3 year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: xinping cao, MD, Principal Investigator — Sun Yat-sen University Cancer Centre
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreu-Martinez FJ, Martinez-Mateu JM. Hypoxia and anaemia in patients with cancer of the uterine cervix. Clin Transl Oncol. 2005 Sep;7(8):323-31. doi: 10.1007/BF02716547. PMID 16185600
- [Background] Timmer PR, Aalders JG, Bouma J. Radical surgery after preoperative intracavitary radiotherapy for Stage IB and IIA carcinoma of the uterine cervix. Gynecol Oncol. 1984 Jun;18(2):206-12. doi: 10.1016/0090-8258(84)90027-1. PMID 6735263
- [Background] Mayr NA, Wen BC, Benda JA, Sorosky JI, Davis CS, Fuller RW, Hussey DH. Postoperative radiation therapy in clinical stage I endometrial cancer: corpus, cervical, and lower uterine segment involvement--patterns of failure. Radiology. 1995 Aug;196(2):323-8. doi: 10.1148/radiology.196.2.7617840.
- [Background] Look KY, Rocereto TF. Relapse patterns in FIGO stage IB carcinoma of the cervix. Gynecol Oncol. 1990 Jul;38(1):114-20. doi: 10.1016/0090-8258(90)90021-c. PMID 2354816
- [Background] Potter ME, Alvarez RD, Shingleton HM, Soong SJ, Hatch KD. Early invasive cervical cancer with pelvic lymph node involvement: to complete or not to complete radical hysterectomy? Gynecol Oncol. 1990 Apr;37(1):78-81. doi: 10.1016/0090-8258(90)90312-9. PMID 2323617
- [Background] Anthopoulos AP, Manetta A, Larson JE, Podczaski ES, Bartholomew MJ, Mortel R. Pelvic exenteration: a morbidity and mortality analysis of a seven-year experience. Gynecol Oncol. 1989 Nov;35(2):219-23. doi: 10.1016/0090-8258(89)90047-4. PMID 2807013